CLINICAL TRIAL: NCT01315938
Title: Abatacept Treatment in Polymyositis and Dermatomyositis
Acronym: ARTEMIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Institute of Rheumatology, Prague (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Ingrid E. Lundberg, Professor, Karolinska Institutet
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-015957-20
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Polymyositis; Dermatomyositis
MeSH Terms: conditions — Polymyositis; Dermatomyositis | interventions — Abatacept

STUDY DESIGN:
Intervention Model Description: Delayed start design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Other): Abatacept will be administered intravenously at a dose based on body weight at the screening visit (baseline): participants weighing <60 kg received 500 mg, 60-100 kg received 750 mg and those >100 kg received 1000 mg.
  Interventions: Drug: Abatacept Active Treatment
- Delayed-onset treatment (Other): Abatacept will be administered intravenously at a dose based on body weight at 3 months: participants weighing <60 kg received 500 mg, 60-100 kg received 750 mg and those >100 kg received 1000 mg.
  Interventions: Drug: Abatacept Delayed-Onset Treatment

INTERVENTIONS:
Drug: Abatacept Active Treatment — Participants will be treated with abatacept by intravenous infusions a total of seven times at week(s) 0, 2, 4, 8, 12, 16 and 20 weeks.
  Other Names: Orencia
  Arms: Active treatment
Drug: Abatacept Delayed-Onset Treatment — Participants will be treated with abatacept for 6 months and received a total of seven intravenous infusions at weeks 12, 14, 16, 20, 24, 28 and 32.
  Other Names: Orencia
  Arms: Delayed-onset treatment

SUMMARY:
The aim of this study is to investigate the efficacy and safety of abatacept in patients with Dermatomyositis (DM) and polymyositis (PM) refractory to conventional treatment using a randomised trial design with delayed start in one arm. Abatacept will be administered intravenously to participants at a dose based on body weight at the screening visit followed by six follow-up treatments (Active treatment arm). Abatacept will also be administered intravenously to participants at a dose based on body weight starting at 3 months followed by six follow-up treatments (Delayed-onset treatment arm). The International Myositis Assessment and Clinical Studies Group (IMACS) preliminary definition of improvement (DOI) will be used for assessment.

DETAILED DESCRIPTION:
This is a phase IIb pilot study with a randomised delayed treatment design. Half of the patients will be randomised to treatment with abatacept from week 0 (Active treatment arm) and half to start active treatment after 3 months (Delayed-onset treatment arm). The open-label study will not include placebo, but the efficacy outcome assessors will be blinded to treatment arm. The study will be conducted at three sites (Karolinska University Hospital Stockholm, Sweden; King's College Hospital National Health Service (NHS), London, United Kingdom (UK); and the Institute of Rheumatology Prague, Prague, Czech Republic).

Patients will be eligible between ages 18 and 80 years and must have active disease after treatment with glucocorticoids (≥0.5 mg/kg/day for ≥1 month), in combination with at least one other immunosuppressive drug, methotrexate (minimum dose 15 mg/week) or azathioprine (minimum dose 100 mg/day) for at least 3 months. Concomitant methotrexate or azathioprine will be allowed, with stable doses for ≥1 month prior to inclusion in the study. Active disease is defined as persisting or worsening muscle weakness (Manual Muscle Test (MMT)-8 bilaterally <150) or low endurance measured by Functional Index for myositis (FI-2) <20% of upper value,15 together with at least one other sign of active disease: elevated (above upper limit of normal) serum levels of muscle enzymes, inflammation in a recent muscle biopsy (<1 month) or on Magnetic resonance imaging (MRI) findings consistent with inflammation, or active extramuscular disease.

The primary endpoint will be the number of responders, defined according to the International Myositis Assessment and Clinical Studies Group (IMACS) preliminary definition of improvement (DOI),16 after treatment with abatacept for 6 months. IMACS DOI is defined as relative improvement by ≥20% in three of any six core set measures, with no more than two core set measures worsening by ≥25%, which cannot be MMT.

Secondary objectives will include the number of responders in the delayed-onset arm compared with active treatment arm at 3 and 6 months, and the change in individual components of the IMACS core set measures for disease activity and in the muscle endurance as tested by FI-2, in the delayed-onset arm compared with active treatment arm at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with definite or probable polymyositis or dermatomyositis diagnosed according to the diagnostic criteria by Bohan and Peter (30,31).
2. For polymyositis a muscle biopsy is required that confirmed this disease (performed at any time before the start of the study) and to exclude other conditions unless a patient is positive for myositis specific or myositis associated autoantibodies.
3. Polymyositis will be included after a judicial process by the three PIs.
4. Inflammatory active disease based on persisting or worsening muscle weakness, MMT < 150 or low endurance, FI -2 < 20% of upper value together with at least one other sign of active disease: elevated serum levels of muscle enzymes (CK, LD, ASAT, ALAT, above upper limit and being explained by muscle involvement and not eg liver disease), inflammation in recent muscle biopsy (< 3 months) or on MRI scans or active extramuscular disease: skin rash, arthritis or interstitial lung disease (ILD) (as suggested by chest X-ray, high resolution computerized tomography (HRCT), or pulmonary function test).
5. Persisting disease activity after a minimum of 3 months treatment with prednisolone or equal drug. The treatment with prednisolone (or equal) should include the dose of at least 0.5 mg/kg/day for at least 1 month in the history and should be stable 1 month prior the baseline visit. Maximum dose of glucocorticoids should not exceed the equivalent of Prednisone 30 mg per day at the time of randomisation.
6. Combination with at least one other immunosuppressive drug, which includes methotrexate (minimum dose 15 mg/week) or azathioprine (minimum dose 100 mg/day) for at least 3 months. The dose of methotrexate or azathioprine should be stable for at least 1 month before the first administration of abatacept.
7. If methotrexate or azathioprine has had to be stopped or the dose decreased due to documented intolerance, lower dose or absence of these drugs is accepted provided this situation is stable for 1 month before the baseline.
8. Age between 18 - 80 years.
9. Signed informed consent.

   -

Exclusion Criteria:

1. Patients with other types of inflammatory myopathies including

   * Drug induced myositis.
   * Inclusion body myositis
   * Malignancy associated myositis.
2. Women who are pregnant or breastfeeding.
3. Women with a positive pregnancy test on enrolment or prior to start of study drug administration.
4. Women of Child Bearing age who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for 10 weeks after the last infusion of study medication.
5. Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, neurological, ophthalmologic or cerebral disease with the exception of those symptoms that are a manifestation of polymyositis or dermatomyositis. Concomitant medical conditions that in the opinion of the investigator might place the subject at unacceptable risk for participation in this study.
6. Subjects with a history of cancer within the last five years (other than non-melanoma skin cell cancers cured by local resection). Existing non-melanoma skin cell cancers must be removed prior to dosing. Patients with dermatomyositis need to be screened for malignancies according to routine procedures.
7. Subjects who have a history of clinically significant drug or alcohol abuse. Subjects currently taking methotrexate who admit to consumption of more than an average of 1 alcoholic drink per day.
8. Subjects with any serious bacterial infection (such as pneumonia, other renal infection and sinusitis), unless treated and resolved with antibiotics or chronic bacterial infection (such as pyelonephritis and chest infection with bronchiectasis) in the previous 3 months.
9. Subjects with active tuberculosis requiring treatment within the previous 3 years. Subjects with a positive PPD at screening will not be eligible for the study unless they completed treatment for latent TB and have a negative chest x-ray at enrolment. A PPD response that is equal to or greater than 10 mm should be considered a positive test, although more conservative criteria may be applied as determined by the clinical circumstance and investigator according to published guidelines and/or local standards endorsed by the medical society. Quantiferon assay may replace PPD testing and patients are excluded from the study if the test is positive. Quantiferon positive patients who completed treatment for latent tuberculosis according to the local guidelines may be considered for enrolment.
10. Subjects with herpes zoster that resolved less than 2 months prior to enrolment.
11. Subjects with evidence (as assessed by the Investigator) of active or latent bacterial or viral infections at the time of potential enrolment, including subjects with evidence of Human Immunodeficiency Virus (HIV) infection.
12. Significant toxicities associated with concomitant or previous immunosuppressive Therapy and anti-TNF therapy that would preclude subjects from participating and completing the study
13. Patients with clinically apparent immunodeficiency syndrome, (IgA deficiency alone is not an exclusion criterion)
14. Subjects with any of the following laboratory values:

    * Hgb < 8.5 g/dL.
    * WBC < 3,000/mm3 (3 x 109/L).
    * Platelets < 100,000/mm3 (100 x 109/L).
    * Serum creatinine > 2 times upper limit of normal.
    * Any other laboratory test results that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study.
15. Subjects previously treated with rituximab: B cell levels are less than lower limit of normal as measured by Fluorescent Activated Cell Sorting (FACS) analysis.
16. For all patients who have received prior rituximab, a normal CD19 B cell count must be documented at the time of screening for this study.
17. Patients with Large granular lymphocyte (LGL) syndrome (to minimize the risk of including patients with high frequency of CD28 null T cells) that may not benefit from treatment.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-11-28 (Actual); Study Completion 2013-11-28 (Actual)

PRIMARY OUTCOMES:
Change in International Myositis Assessment and Clinical Studies Group (IMACS) | Change from Baseline IMACS at 6 months
  The primary endpoint will be the number of responders, defined according to the International Myositis Assessment and Clinical Studies Group (IMACS) preliminary definition of improvement (DOI) after treatment with abatacept for 6 months. IMACS DOI is defined as relative improvement by ≥20% in three of any six core set measures, with no more than two core set measures worsening by ≥25%, which cannot be MMT.

SECONDARY OUTCOMES:
Change in International Myositis Assessment and Clinical Studies Group (IMACS) | Change from 3 IMACS at 6 months
  The number of responders in the delayed-onset arm compared with active treatment arm at 3 and 6 months, and the change in individual components of the IMACS core set measures for disease activity and in the muscle endurance as tested by FI-2, in the delayed-onset arm compared with active treatment arm at 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid E Lundberg, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Institute of Rheumatology, Prague, Czechia
- Karolinska University Hospital, Stockholm, Sweden